CLINICAL TRIAL: NCT00297856
Title: Open, Prospective Study of the Safety of GSK Biologicals' Boostrix® (Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine, Adsorbed) Administered to a Cohort of Adolescents in a US Health Maintenance Organization (HMO)
Brief Title: Post-marketing Safety Study of GSK Biologicals' Boostrix® Vaccine
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 104154
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Diphtheria; Tetanus; Acellular Pertussis
Keywords: Boostrix
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Boostrix; Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Boostrix cohort
  Interventions: Biological: Boostrix®
- Historical Td cohort
  Interventions: Biological: Td (Tetanus diphtheria) vaccine

INTERVENTIONS:
Biological: Boostrix® — Single dose
  Groups: Boostrix cohort
Biological: Td (Tetanus diphtheria) vaccine — Single dose
  Groups: Historical Td cohort

SUMMARY:
Pre-licensure studies of GSK Biologicals' Boostrix® have shown it to be generally safe and well-tolerated. This post-licensure study is designed to evaluate relatively uncommon/rare outcomes in a large population cohort. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Data collection through utilization of automated databases at the study site. The collaborator is Kaiser Permanente Vaccine Study Center.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the age of 10 and 18 years (inclusive) who received a dose of Boostrix and who have safety follow-up information available

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects enrolled in the Northern California Kaiser-Permanente Health Care Plan
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of medically-attended neurological events. | 30 days following vaccination with Boostrix.

SECONDARY OUTCOMES:
Occurrence of medically-attended hematologic events | 30 days following vaccination with Boostrix
Occurrence of allergic reactions. | 30 days following vaccination with Boostrix
Occurrence of new onset chronic illnesses | 6-month period following vaccination with Boostrix
Occurrence of neurological and hematological events and allergic reactions | Within the second 30-day period following vaccination with Boostrix
Occurrence of chronic illnesses in an historical control cohort of subjects vaccinated with Td vaccine

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Oakland, California, United States

REFERENCES:
- [Background] Klein NP, Hansen J, Lewis E, Lyon L, Nguyen B, Black S, Weston WM, Wu S, Li P, Howe B, Friedland LR. Post-marketing safety evaluation of a tetanus toxoid, reduced diphtheria toxoid and 3-component acellular pertussis vaccine administered to a cohort of adolescents in a United States health maintenance organization. Pediatr Infect Dis J. 2010 Jul;29(7):613-7. doi: 10.1097/INF.0b013e3181d581f9. PMID 20190673